CLINICAL TRIAL: NCT03670459
Title: Cawthorne Cooksey Versus Vestibular Habituation Exercises on Trunk Kinetics and Velocity of Gait in Patients With Multiple Sclerosis
Brief Title: Forty Five Patients With Multiple Sclerosis Recieved Vestibular Rehabilitation and Balance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Hosam Magdy Metwally, Hossam.magdy.pt@o6u.edu.eg, October 6 University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Identifier No. 11
Record Dates: First submitted 2018-09-07; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Neurologic Disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Patients in G1 will receive traditional physical therapy program (balance exercises) for twelve sessions; day after day
  Interventions: Other: Balance exercises
- Group 2 (Experimental): Patients in G2 will receive Cawthorne Cooksey Exercises in addition to traditional physical therapy program for twelve sessions; day after day .
  Interventions: Other: Cawthorne Cooksey exercises
- Group 3 (Experimental): Patients in G3 will receive vestibular habituation exercises in addition to traditional physical therapy program for twelve sessions; day after day.
  Interventions: Other: Vestibular habituation exercises

INTERVENTIONS:
Other: Cawthorne Cooksey exercises — Eye movements and head movements
  Arms: Group 2
Other: Vestibular habituation exercises — Move from a sitting position to flat on the back
  Arms: Group 3
Other: Balance exercises — Weight Shift Forward and Back
  Arms: Group 1

SUMMARY:
Patients with multiple sclerosis (MS) might develop dizziness or vertigo as a first manifestation or during the course of the illness. Many patients with MS experience chronic or intermittent dizziness. Acute symptoms of dizziness or vertigo in MS fall into two categories; acute vestibular syndrome (AVS) and positional vertigo.

Vestibular disorder due to MS decreases whole body dynamic postural control and causes many functional limitations as limitations in ambulation, dynamic balance and trunk control and that decreases the quality of life.

Vestibular dysfunction has long been recognized as causing some of the most common symptoms in MS, true vertigo is found at presentation in up to 17% of patients, several recent reports have suggested that vestibular symptoms develop early in the disease process. Vestibular Rehabilitation has been shown to be effective in reducing symptoms and improving function for patients with vestibular disorders. The goal of vestibular rehabilitation is to promote the central nervous system compensation through exercise-based strategies.

DETAILED DESCRIPTION:
The purposes of the study were to:

* Measure the effect of Cawthorne Cooksey Exercises on trunk kinetics and velocity of gait in patient with MS.
* Measure the effect of vestibular habituation on trunk kinetics and velocity of gait in patient with MS.
* Determine which type of vestibular exercises had more effect on the rehabilitation of patients with MS Cawthorne Cooksey or vestibular habituation?
* Determine if there was a correlation between the improvement in trunk kinetics and velocity of gait in patients with MS.

Forty five patients with multiple sclerosis were selected from the Out Patient Clinics of Neurology and Internal Medicine in Kasr Al- Aini Hospitals, Out Patient Clinic of Neurology, Faculty of Physical Therapy, Cairo University and 6th of October central hospital.

The selected patients were divided into three equal groups:

* Patients in G1 will receive traditional physical therapy program (balance training) for twelve sessions; day after day
* Patients in G2 will receive Cawthorne Cooksey Exercises in addition to traditional physical therapy program for twelve sessions; day after day.
* Patients in G3 will receive vestibular habituation exercises in addition to traditional physical therapy program for twelve sessions; day after day.

ELIGIBILITY:
Inclusion Criteria:

* All the Patients in this study will be referred from the neurologist and will be diagnosed as relapsing-remitting multiple sclerosis in the form of hemiparesis with muscle tone of 1,1+ modified Ashworth scale.
* The diagnosis will be confirmed by MRI or CT scan and all the patients will follow the neurological examination.
* Forty five female patients ages will range from 35-55 years.
* All selected patients with central vertigo (central vestibular disorder) according to Dix Hallpike test (Cohen, 2004)
* The Degree of disability of multiple sclerosis will be from 2 - 2.5 (according to expanded disability status scale (EDSS)) (Kaufman et al, 2000)
* All the selected patients will have grade 3 group muscle test of lower limb muscles.
* All the selected patients will have scored 27-30 in mini-mental state examination (Crum et al, 1993)
* Patients who are selected in the study will be ambulant.
* Patients will be medically stable.

Exclusion Criteria:

* Patients with musculoskeletal deformity.
* Patients with diabetes mellitus.
* Patients with psychological disturbance or seizures.
* Patients with visual or impairment.
* Patients with inner ear disorders
* Patients with other neurological disorders such as cerebellar lesion

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-12-31 (Actual); Primary Completion 2018-07-21 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Isokinetic dynamometer | up to 30 days
  Assessment of trunk kinetics

CONTACTS AND LOCATIONS:
Overall Officials: Hosam Magdy Metwally, Doctoral, Principal Investigator — October 6 University
Locations (1):
- October 6 University, Giza, Egypt